CLINICAL TRIAL: NCT04487769
Title: Early Lung Ultrasound Score Predicts Duration of Ventilation and ICU Mortality in COVID-19 Invasively Ventilated Patients
Brief Title: Lung Ultrasound in COVID-19 Patients
Acronym: LUS-COVID
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Centre Hospitalier Universitaire de Brussels, Brussels, Belgium (Unknown); Miulli Regional Hospital, Acquaviva delle Fonti, Italy (Unknown); University of Foggia (Other); University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. M.J. Schultz, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: LUS-COVID
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Covid19; Ultrasound; ARDS
Keywords: new coronavirus disease; coronavirus disease 2019; lung imaging; lung ultrasound; lung ultrasound score; prognostication; duration of ventilation; mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the prognostic performance of an early global LUS score with respect to the mortality in ICU and duration of ventilation.

DETAILED DESCRIPTION:
This is an international multicenter cohort study on data collected between March and April 2020. The first available lung ultrasound examination that used a 12-regions approach was used to calculate the global LUS score.

Patients are included if they fulfilled the following criteria: 1) admitted to one of the participating ICU; 2) for invasive ventilation; 3) for respiratory failure due to confirmed COVID-19; and 4) having had a LUS examination performed within the first week of start of invasive ventilation.

The primary and secondary outcomes were liberation from invasive ventilation and mortality.

Demographic, clinical and outcome variables will be presented as percentages for categorical variables and as medians with interquartile ranges (IQR) for continuous variables.

Receiver operating characteristics (ROC) analysis will be used to derive the prognostic discriminatory performance of global LUS score in determining succesful extubation and mortality at day 28. The Youden index will be used to derive the optimal cut-off. The association of global LUS with unfavourable outcomes are analyzed with Cox proportional hazard analysis (for successful extubation and alive at day 28), logistic regression models (mortality at day 28). Hazard ratio or odds ratio with 95% confidence intervals were calculated for each outcome.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an ICU participating in this study between February 1, 2020 and April 30, 2020
* Confirmed with reverse transcriptase polymerase chain reaction (RT-PCR) COVID-19 infection
* Having had received invasive ventilation
* Having had examined at least once with lung ultrasound under invasive ventilation

Exclusion Criteria:

* Age <18 years
* First examination with LUS in patients already under extracorporeal membrane oxygenation (ECMO) support.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe COVID-19 infection under invasive ventilation who received lung ultrasound examination as a standard care.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Liberation from invasive ventilation | 28 days
  Patient who survived but remained invasively ventilated up to day 28 were marked without event. Patients who survived but were extubated were marked with an event at the day of successful extubation.

SECONDARY OUTCOMES:
Mortality | 28 days
  Patient who survived up to day 28 were marked without event. Patients who survived but were extubated were marked with an event at the day of successful extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, MD, Principal Investigator — Amsterdam University Medical Centers, location 'AMC'
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pierrakos C, Lieveld A, Pisani L, Smit MR, Heldeweg M, Hagens LA, Smit J, Haaksma M, Veldhuis L, Schmidt RW, Errico G, Marinelli V, Attou R, David CE, Zimatore C, Murgolo F, Grasso S, Mirabella L, Cinnella G, De Bels D, Schultz MJ, Tuinman PR, Bos LD. A Lower Global Lung Ultrasound Score Is Associated with Higher Likelihood of Successful Extubation in Invasively Ventilated COVID-19 Patients. Am J Trop Med Hyg. 2021 Oct 18;105(6):1490-1497. doi: 10.4269/ajtmh.21-0545. PMID 34662857